CLINICAL TRIAL: NCT04147650
Title: A Randomized, Double-Masked, Vehicle-Controlled, Dose Ranging Study to Assess the Efficacy and Safety of Voclosporin Ophthalmic Solution (VOS) in Subjects With Dry Eye Syndrome (DES)
Brief Title: Dose Ranging Study to Assess the Efficacy and Safety of Voclosporin Ophthalmic Solution in Subjects With Dry Eye Syndrome
Acronym: AUDREY
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Aurinia Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AUR-VOS-2019-01
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Results first posted 2021-12-10 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Dry Eye Syndrome; Keratoconjunctivitis Sicca
Keywords: Dry Eye Calcineurin Inhibitors; Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to one of the following treatment groups:
  Investigational product (IP): one drop 0.05% VOS, in both eyes (OU) twice a day (BID) over 12 weeks, one drop 0.10% VOS OU BID over 12 weeks, or one drop 0.20% VOS OU BID over 12 weeks.
  Comparator: one drop VOS vehicle OU BID over 12 weeks.
Who Masked: Participant, Investigator
Masking Description: Double masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 0.05% Voclosporin Ophthalmic Solution (VOS) (Experimental): 0.05% VOS, in both eyes (OU) twice a day (BID) over 12 weeks
  Interventions: Drug: 0.05% Voclosporin Ophthalmic Solution (VOS)
- 0.10% VOS (Experimental): 0.10% VOS, in both eyes (OU) twice a day (BID) over 12 weeks
  Interventions: Drug: 0.10% VOS
- 0.20% VOS (Experimental): 0.20% VOS, in both eyes (OU) twice a day (BID) over 12 weeks
  Interventions: Drug: 0.20% VOS
- Vehicle Ophthalmic Solution (Placebo Comparator): Vehicle Ophthalmic Solution, in both eyes (OU) twice a day (BID) over 12 weeks
  Interventions: Drug: Vehicle Ophthalmic Solution

INTERVENTIONS:
Drug: 0.05% Voclosporin Ophthalmic Solution (VOS) — 0.05% VOS, in both eyes (OU) twice a day (BID) over 12 weeks
  Arms: 0.05% Voclosporin Ophthalmic Solution (VOS)
Drug: 0.10% VOS — 0.10% VOS, in both eyes (OU) twice a day (BID) over 12 weeks
  Arms: 0.10% VOS
Drug: 0.20% VOS — 0.20% VOS, in both eyes (OU) twice a day (BID) over 12 weeks
  Arms: 0.20% VOS
Drug: Vehicle Ophthalmic Solution — Vehicle Ophthalmic Solution, in both eyes (OU) twice a day (BID) over 12 weeks
  Arms: Vehicle Ophthalmic Solution

SUMMARY:
A Multi-Center, Phase 2/3, Randomized, Double-Masked, Parallel-Group, Vehicle-Controlled, Clinical Trial to Assess the Safety and Efficacy of Voclosporin Ophthalmic Solution (0.05%, 0.10%, 0.20%) Compared to Vehicle in Subjects with Dry Eye Syndrome.

DETAILED DESCRIPTION:
This is a Phase 2/3, multi-center, randomized, double-masked, vehicle-controlled study to assess the efficacy and safety of three different concentrations of VOS when administered in both eyes (OU) twice a day (BID) over 12 weeks in subjects with mild to moderate DES. Subjects will undergo a 14- to 17-day run-in period in which VOS vehicle will be self-administered OU, BID. Subjects will be re-assessed to confirm they meet all of the inclusion criteria and none of the exclusion criteria. It is estimated that the study will enroll approximately 480 subjects across approximately 9 study centers. Eligible subjects will be randomized in a 1:1:1:1 ratio to one of the following study treatment groups after the 14- to 17-day run-in period.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age.
* Have a documented history of Dry Eye prior to Visit 1.
* Willing and able to follow protocol procedures and instructions.

Exclusion criteria:

* Have undergone cataract or LASIK surgery within 1 year prior to Visit 1.
* Recent or current evidence of infection or inflammation in either eye.
* Current evidence of blepharitis, other meibomian gland dysfunction, conjunctivitis or history of herpes simplex or zoster keratitis in either eye.
* Have used any investigational drug or device within 30 days prior to Visit 1.
* Have used ophthalmic drugs (any topical eye medications) including prescription medication and over the counter (OTC) agents on the date of Visit 1.
* Have worn contact lenses 24 hours prior to Visit 1.
* Have used Xiidra® (lifitegrast) within 14 days prior to Visit 1.
* Have used Calcineurin Inhibitors (CNIs) such as Restasis® (cyclosporin ophthalmic emulsion) or CequaTM within 30 days prior to Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2020-09-17 (Actual); Study Completion 2020-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Palmen, Study Director — Aurinia Pharmaceuticals
Locations (9):
- United States (9):
  - Aurinia Investigative Center, Newport Beach, California
  - Aurinia Investigative Center, Colorado Springs, Colorado
  - Aurinia Investigative Center, Louisville, Kentucky
  - Aurinia Investigative Center, Lewiston, Maine
  - Aurinia Investigative Center, Andover, Massachusetts
  - Aurinia Investigative Center, Raynham, Massachusetts
  - Aurinia Investigative Center, Cranberry Township, Pennsylvania
  - Aurinia Investigative Center, Memphis, Tennessee
  - Aurinia Investigative Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 0.05% Voclosporin Ophthalmic Solution (VOS) | 0.10% VOS | 0.20% VOS | Vehicle Ophthalmic Solution
Started | 127 | 126 | 128 | 127
Modified Intent to Treat (mITT) | 120 | 119 | 122 | 121
Completed | 116 | 107 | 121 | 120
Not Completed | 11 | 19 | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.05% Voclosporin Ophthalmic Solution (VOS) | 0.10% VOS | 0.20% VOS | Vehicle Ophthalmic Solution | Total
Number analyzed (Participants) | 127 | 126 | 128 | 127 | 508
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (11.82) | 64.2 (11.27) | 64.8 (10.47) | 64.1 (12.43) | 64.1 (11.49)
Age, Continuous [Median (Full Range); unit: years] | 64 [25 to 86] | 65 [30 to 84] | 65 [28 to 89] | 65 [27 to 94] | 65 [25 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 91 | 88 | 97 | 372
  Male | 31 | 35 | 40 | 30 | 136
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 7 | 6 | 25
  Not Hispanic or Latino | 120 | 120 | 121 | 121 | 482
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 0 | 1 | 4
  Asian | 7 | 5 | 9 | 10 | 31
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1 | 2
  Black or African American | 17 | 16 | 17 | 22 | 72
  White | 96 | 103 | 99 | 91 | 389
  More than one race | 4 | 1 | 3 | 2 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With a ≥10 mm Increase From Baseline in Schirmer Tear Test (STT)
Description: Number of subjects with a ≥10 mm increase from baseline in STT at Week 4 in the study eye. The STT scale is a measure of tear production with a minimum of 0 mm and no there is no specified maximum for this scale.
Time Frame: 4 Weeks
Population: Modified intent to treat (mITT) number of subjects achieving ≥10 mm increase improvement at week 4
Measure: Number; unit: participants
Arm/Group | 0.05% Voclosporin Ophthalmic Solution (VOS) | 0.10% VOS | 0.20% VOS | Vehicle Ophthalmic Solution
Number analyzed (Participants) | 120 | 119 | 122 | 121
participants | 12 | 10 | 13 | 6
Statistical Analysis 1: Comparison: 0.05% Voclosporin Ophthalmic Solution (VOS); 0.05 % VOS versus vehicle; Test type: Superiority; p = 0.1352, Regression, Logistic; Odds Ratio (OR) = 2.18, 95% CI 2-sided [0.62 to 7.62]
Statistical Analysis 2: Comparison: 0.10% VOS; 0.10% VOS versus vehicle; Test type: Superiority; p = 0.2823, Regression, Logistic; Odds Ratio (OR) = 1.78, 95% CI 2-sided [0.49 to 6.45]
Statistical Analysis 3: Comparison: 0.20% VOS; 0.20% VOS versus vehicle; Test type: Superiority; p = 0.0889, Regression, Logistic; Odds Ratio (OR) = 2.41, 95% CI 2-sided [0.70 to 8.30]

2. Secondary Outcome: Change From Baseline in Eye Dryness
Description: Mean change from baseline in Eye Dryness Visual Analogue Scale (VAS) in subjects with a baseline Eye Dryness VAS score ≥ 60 mm. Eye Dryness Visual Analogue Scale 0-100 mm, where 0 corresponds to "no discomfort" and 100 corresponds to "maximal discomfort."
Time Frame: Value at 4 Weeks minus value at baseline
Population: The analysis was performed using all mITT subjects with a baseline eye dryness VAS ≥60 mm. Subjects without a Week 4 eye dryness VAS score were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 0.05% Voclosporin Ophthalmic Solution (VOS) | 0.10% VOS | 0.20% VOS | Vehicle Ophthalmic Solution
Number analyzed (Participants) | 85 | 84 | 86 | 89
units on a scale | -10.6 (21.80) | -9.3 (20.00) | -5.0 (17.68) | -7.0 (17.59)
Statistical Analysis 1: Comparison: 0.05% Voclosporin Ophthalmic Solution (VOS); 0.05% VOS versus vehicle; Test type: Superiority; p = 0.3604, ANCOVA; Least square mean difference = -2.6, 95% CI 2-sided [-9.6 to 4.3]
Statistical Analysis 2: Comparison: 0.10% VOS; 0.10% VOS versus vehicle; Test type: Superiority; p = 0.3737, ANCOVA; Least square mean difference = -2.6, 95% CI 2-sided [-9.6 to 4.4]
Statistical Analysis 3: Comparison: 0.20% VOS; 0.20% VOS versus vehicle; Test type: Superiority; p = 0.5307, ANCOVA; Least square mean difference = 1.8, 95% CI 2-sided [-5.1 to 8.6]

ADVERSE EVENTS:
Time Frame: Day 1 to Week 13
Arm/Group | 0.05% Voclosporin Ophthalmic Solution (VOS) | 0.10% VOS | 0.20% VOS | Vehicle Ophthalmic Solution
All-Cause Mortality (participants affected / at risk) | 0/127 | 1/126 | 0/128 | 0/127
Serious Adverse Events (participants affected / at risk) | 1/127 | 3/126 | 2/128 | 3/127
Other Adverse Events (participants affected / at risk) | 29/127 | 42/126 | 44/128 | 8/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.05% Voclosporin Ophthalmic Solution (VOS) (N=127) | 0.10% VOS (N=126) | 0.20% VOS (N=128) | Vehicle Ophthalmic Solution (N=127)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.05% Voclosporin Ophthalmic Solution (VOS) (N=127) | 0.10% VOS (N=126) | 0.20% VOS (N=128) | Vehicle Ophthalmic Solution (N=127)
Instillation site pain (General disorders) | 29 (30) | 42 (43) | 44 (47) | 8 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (4):
  • Study Protocol: Version 1.0 (2019-07-26): https://cdn.clinicaltrials.gov/large-docs/50/NCT04147650/Prot_000.pdf
  • Study Protocol: Version 2.0 (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/50/NCT04147650/Prot_001.pdf
  • Study Protocol: Version 3.0 (2020-06-26): https://cdn.clinicaltrials.gov/large-docs/50/NCT04147650/Prot_002.pdf
  • Statistical Analysis Plan (2020-06-26): https://cdn.clinicaltrials.gov/large-docs/50/NCT04147650/SAP_003.pdf